CLINICAL TRIAL: NCT00240253
Title: A Randomized, Double-Blind, Placebo-Controlled, Multicenter Study Evaluating the Efficacy and Safety of Adding Symlin® to Lantus® (Insulin Glargine) in Subjects With Type 2 Diabetes Who Are Not Achieving Glycemic Targets
Brief Title: A Study Evaluating the Efficacy and Safety of Adding Symlin® to Lantus® (Insulin Glargine) in Subjects With Type 2 Diabetes
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 137-156
Record Dates: First submitted 2005-10-14; First posted 2005-10-18 (Estimated); Last update posted 2015-03-31 (Estimated); Status verified 2015-03

CONDITIONS: Type 2 Diabetes Mellitus
Keywords: diabetes; Amylin; Symlin; pramlintide; insulin glargine
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Diabetes Mellitus | interventions — pramlintide

ARMS (1):
- Pramlintide (Active Comparator)
  Interventions: Drug: pramlintide acetate

INTERVENTIONS:
Drug: pramlintide acetate — Clear, colorless, sterile solution for SC injection

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of adding Symlin to an established regimen of insulin glargine in subjects with type 2 diabetes who are not achieving glycemic targets.

ELIGIBILITY:
Inclusion Criteria:

* Has HbA1c >7.0% and <=10.5%
* Has a body mass index (BMI) >=25 kg/m2 and <=45 kg/m2
* Has received insulin glargine for 3 months prior to study start and has been on a stable dose for 1 month prior to study start
* If taking oral antidiabetic agents, has been on a stable dose for at least 2 months

Exclusion Criteria:

* Has been previously treated with Symlin/pramlintide (or has participated in a Symlin/pramlintide clinical study)
* Has received any investigational drug within 1 month of screening

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2005-10; Primary Completion 2006-06 (Actual); Study Completion 2006-06 (Actual)

PRIMARY OUTCOMES:
To evaluate the efficacy and safety of adding Symlin to an established regimen of insulin glargine in subjects with type 2 diabetes. | 16 Weeks

SECONDARY OUTCOMES:
To evaluate the effects of adding Symlin to an established regimen of insulin glargine in subjects with type 2 diabetes on markers of cardiovascular risk, fasting serum lipids, fasting plasma glucose, waist circumference, and patient-reported outcomes. | 16 Weeks

CONTACTS AND LOCATIONS:
Overall Officials: Lisa Porter, MD, Study Director — Amylin Pharmaceuticals, LLC.
Locations (34):
- United States (34):
  - Research Site, Phoenix, Arizona
  - Research Site, Concord, California
  - Research Site, La Jolla, California
  - Research Site, Los Gatos, California
  - Research Site, Salinas, California
  - Research Site, Walnut Creek, California
  - Research Site, Denver, Colorado
  - Research Site, New Britain, Connecticut
  - Research Site, Washington D.C., District of Columbia
  - Research Site, Palm Harbor, Florida
  - Research Site, Atlanta, Georgia
  - Research Site, Indianapolis, Indiana
  - Research Site, Wichita, Kansas
  - Research Site, Lexington, Kentucky
  - Research Site, Baton Rouge, Louisiana
  - Research Site, Bloomfield Hills, Michigan
  - Research Site, Detroit, Michigan
  - Research Site, Grand Rapids, Michigan
  - Research Site, Chesterfield, Missouri
  - Research Site, Butte, Montana
  - Research Site, Omaha, Nebraska
  - Research Site, Charlotte, North Carolina
  - Research Site, Durham, North Carolina
  - Research Site, Cincinnati, Ohio
  - Research Site, Oklahoma City, Oklahoma
  - Research Site, Medford, Oregon
  - Research Site, Portland, Oregon
  - Research Site, Philadelphia, Pennsylvania
  - Research Site, Tipton, Pennsylvania
  - Research Site, Nashville, Tennessee
  - Research Site, Dallas, Texas
  - Research Site, Charlottesville, Virginia
  - Research Site, Olympia, Washington
  - Research Site, Spokane, Washington

REFERENCES:
- [Derived] Peyrot M, Rubin RR, Polonsky WH. Diabetes distress and its association with clinical outcomes in patients with type 2 diabetes treated with pramlintide as an adjunct to insulin therapy. Diabetes Technol Ther. 2008 Dec;10(6):461-6. doi: 10.1089/dia.2008.0031. PMID 19049375
- [Derived] Wysham C, Lush C, Zhang B, Maier H, Wilhelm K. Effect of pramlintide as an adjunct to basal insulin on markers of cardiovascular risk in patients with type 2 diabetes. Curr Med Res Opin. 2008 Jan;24(1):79-85. doi: 10.1185/030079908x253537. PMID 18031595
- [Derived] Riddle M, Frias J, Zhang B, Maier H, Brown C, Lutz K, Kolterman O. Pramlintide improved glycemic control and reduced weight in patients with type 2 diabetes using basal insulin. Diabetes Care. 2007 Nov;30(11):2794-9. doi: 10.2337/dc07-0589. Epub 2007 Aug 13. PMID 17698615